CLINICAL TRIAL: NCT00274989
Title: Multicentre Phase II Trial of Bendamustine in Combination With Rituximab for Patients With Previously Untreated or Relapsed Chronic Lymphocytic Leukemia. CLL2M Protocol of the German CLL-Study Group (GCLLSG)
Brief Title: Bendamustine and Rituximab in Treating Patients With Previously Untreated or Relapsed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2M; EU-20552; ROCHE-GCLLSG-CLL2M; 2005-001596-34 (EudraCT Number)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: B-cell chronic lymphocytic leukemia; relapsed refractory chronic lymphocytic leukemia; previously untreated chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine plus Rituximab (Experimental)
  Interventions: Drug: Bendamustine; Biological: Rituximab

INTERVENTIONS:
Drug: Bendamustine — First-Line Therapy: Bendamustine i.v. 90 mg/m² day 1-2, q4wks, cycle 1 to 6
  2nd to 4th -Line Therapy: Bendamustine i.v. 70 mg/m² day 1-2 q4wks, cycle 1 to 6
Biological: Rituximab — First-Line Therapy: Rituximab i.v. 375 mg/m² day 0, q4wks, cycle 1; Rituximab i.v. 500 mg/m² day 1, q4wks, cycle 2-6
  2nd to 4th -Line Therapy: Rituximab i.v. 375 mg/m² day 0, q4wks, cycle 1; Rituximab i.v. 500 mg/m² day 1, q4wks, cycle 2-6
  Other Names: MabThera, Rituxan

SUMMARY:
CLL2M is a phase 2, multicenter, open label study to investigate the possible therapeutic benefits of using bendamustine in combination with rituximab for the treatment of patients with previously untreated or relapsed CLL.

DETAILED DESCRIPTION:
Conventional chemotherapy and also high dose chemotherapy with autologous stem cell transplantation are not curative treatment options in B-CLL; nearly all patients will eventually relapse. Also monoclonal antibodies are not curative for B-CLL patients in monotherapy, their impact on survival in combination with conventional chemotherapy is currently validated. In addition, there is no standard combination therapy for patients with relapsed CLL. Therefore there is an urgent medical need to identify new strategies.

The combination of rituximab (monoclonal antibody) and bendamustine (chemotherapy) has shown encouraging activity in patients with relapsed/refractory NHL or mantle cell lymphoma. In vitro studies have been used to investigate the effects of bendamustine and rituximab on programmed cell death (apoptosis) and have shown synergistic effects of both drugs. The mechanisms of action of these two active drugs may provide a treatment with good therapeutic potential in CLL. However, though bendamustine has been used for over 30 years there is still a need to define a standard regimen for the use of bendamustine in combination with monoclonal antibodies (mAb) especially in the treatment of CLL.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of B-CLL in need of treatment

  * Previously untreated Binet stage C or Binet B with need of treatment according to NCI-criteria
  * Relapsed or refractory disease after at least one but not more than 3 prior regimens. Patients who previously received bendamustine must have had at least a partial response with duration of response of at least six months.
* World Health Organization performance status of 0-2
* Life expectancy >12 weeks
* Anti-cancer therapy, major surgery, or irradiation was completed >3 weeks before registration in this study. Patient must have recovered from the acute side effects incurred as a result of previous therapy.
* Serum creatinine ≤1.5 the institutional upper limit of normal (ULN) or Creatinine clearance >30 ml/min/1.73 m²
* Adequate liver function as indicated by a total bilirubin, AST, and ALT ≤2 the institutional ULN value, unless directly attributable to the patient's tumor.
* Female patients with childbearing potential must have a negative serum pregnancy test within two weeks of first dose of study drug(s). Male and female patients must agree to use an effective contraceptive method while on study treatment and for a minimum of six months following study therapy.
* Signed, written informed consent.

Exclusion Criteria:

* Previously treated with >3 prior regimens for B-CLL.
* Known central nervous system (CNS) involvement with B-CLL.
* Patients who have progressed with more aggressive B-cell cancers such as Richter's syndrome.
* History of anaphylaxis following exposure to monoclonal antibodies.
* Known to be human immunodeficiency virus (HIV), hepatitis B, or C positive.
* Active infection or history of severe infection (grade 4) within 3 months prior to study registration.
* Medical condition requiring prolonged use of oral corticosteroids (> 1 month).
* Use of investigational agents within 30 days prior to study randomization.
* Active secondary malignancy.
* ANC <1.5x109/L or platelet count <75x109/L, unless due to bone marrow involvement of CLL.
* Other severe, concurrent diseases, including tuberculosis, mental disorders, serious cardiac functional capacity (Class III or IV as defined by the New York Heart Association Classification), severe diabetes, severe hypertension, pulmonary disease (chronic obstructive pulmonary disease [COPD] with hypoxemia), or major organ malfunction (liver, kidney) that could interfere with the patient's ability to participate in the study.
* Pregnant or nursing women.
* Any circumstance at the time of study entry that would preclude completion of the study or the required follow-up.
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2005-11; Primary Completion 2008-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 56 days after the last of six cycles
  Response will be assessed using clinical examination, hematology, bone marrow examination, plain radiograph of the chest (chest X-ray), ultrasound or CT of the abdomen, and MRD testing (for the molecular response rate only).

CONTACTS AND LOCATIONS:
Overall Officials: Clemens M. Wendtner, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (58):
- Germany (58):
  - Internistische Praxis - Arnstadt, Arnstadt
  - Klinikum Augsburg, Augsburg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - Charite - Campus Charite Mitte, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Marienhospital Bottrop gGmbH, Bottrop
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Klinikum Darmstadt, Darmstadt
  - Krankenhaus Benrath, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Universitaetsklinikum Essen, Essen
  - Staedtische Kliniken Esslingen, Esslingen am Neckar
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Internistische Praxisgemeinschaft, Germering
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Allgemeines Krankenhaus Hagen, Hagen
  - Praxis fur Innere Medizin - Hamburg, Hamburg
  - Hamatologische/Onkologische - Hamburg, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Universitaetsklinikum des Saarlandes, Homburg
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Klinikum Lippe - Lemgo, Lemgo
  - Gemeinschaftspraxis - Ludwigshafen, Ludwigshafen
  - Kreiskrankenhaus Luedenscheid, Lüdenscheid
  - Staedtisches Klinikum Magdeburg, Magdeburg
  - Krankenhaus Maria Hilf GmbH, Mönchengladbach
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Haematologisch - Onkologische Gemeinschaftspraxis - Muenster, Münster
  - Onkologische Schwerpunktpraxis Dr. Schmidt, Neunkirchen
  - Klinikum Oldenburg, Oldenburg
  - Paracelsus Karankenhaus Ruit, Ostfildern
  - Gemeinschaftspraxis - Pinneberg, Pinnebeg
  - Klinikum Ernst Von Bergmann, Potsdam
  - Scherpunktpraxis fur Hematologie und Onkologie, Regensburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Internistische Praxis Dres. Hempel und Hochdorfer, Rehling
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Caritasklinik St. Theresia, Saarbrücken
  - Schwerpunktpraxis fur Hamatologie und Onkologie, Siegburg
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Hanse-Klinikum Stralsund - Krankenhaus West, Stralsund
  - Haematologische Praxis, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - St. Marienhospital - Vechta, Vechta
  - Heinrich-Braun-Krankenhaus Zwickau, Zwickau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Sawaf O, Robrecht S, Bahlo J, Fink AM, Cramer P, von Tresckow J, Maurer C, Bergmann M, Seiler T, Lange E, Kneba M, Stilgenbauer S, Dohner H, Kiehl MG, Jager U, Wendtner CM, Fischer K, Goede V, Hallek M, Eichhorst B, Hopfinger G. Impact of gender on outcome after chemoimmunotherapy in patients with chronic lymphocytic leukemia: a meta-analysis by the German CLL study group. Leukemia. 2017 Oct;31(10):2251-2253. doi: 10.1038/leu.2017.221. Epub 2017 Jul 12. No abstract available. PMID 28745332
- [Background] Sachanas S, Pangalis GA, Fink AM, Bahlo J, Fischer K, Levidou G, Kyrtsonis MC, Bartzi V, Vassilakopoulos TP, Kalpadakis C, Koulieris E, Moschogiannis M, Yiakoumis X, Tsirkinidis P, Angelopoulou MK, Eichhorst B, Hallek M. Small Lymphocytic Lymphoma: Analysis of Two Cohorts Including Patients in Clinical Trials of the German Chronic Lymphocytic Leukemia Study Group (GCLLSG) or in "Real-Life" Outside of Clinical Trials. Anticancer Res. 2019 May;39(5):2591-2598. doi: 10.21873/anticanres.13382. PMID 31092457
- [Result] Fischer K, Cramer P, Busch R, Stilgenbauer S, Bahlo J, Schweighofer CD, Bottcher S, Staib P, Kiehl M, Eckart MJ, Kranz G, Goede V, Elter T, Buhler A, Winkler D, Kneba M, Dohner H, Eichhorst BF, Hallek M, Wendtner CM. Bendamustine combined with rituximab in patients with relapsed and/or refractory chronic lymphocytic leukemia: a multicenter phase II trial of the German Chronic Lymphocytic Leukemia Study Group. J Clin Oncol. 2011 Sep 10;29(26):3559-66. doi: 10.1200/JCO.2010.33.8061. Epub 2011 Aug 15. PMID 21844497
- [Result] Fischer K, Cramer P, Busch R, Bottcher S, Bahlo J, Schubert J, Pfluger KH, Schott S, Goede V, Isfort S, von Tresckow J, Fink AM, Buhler A, Winkler D, Kreuzer KA, Staib P, Ritgen M, Kneba M, Dohner H, Eichhorst BF, Hallek M, Stilgenbauer S, Wendtner CM. Bendamustine in combination with rituximab for previously untreated patients with chronic lymphocytic leukemia: a multicenter phase II trial of the German Chronic Lymphocytic Leukemia Study Group. J Clin Oncol. 2012 Sep 10;30(26):3209-16. doi: 10.1200/JCO.2011.39.2688. Epub 2012 Aug 6. PMID 22869884